CLINICAL TRIAL: NCT03947177
Title: Culturally Enhancing a Motivational Interviewing Intervention For Latinx Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Virginia Foundation of Healthy Youth (Unknown); Sacred Heart Center (Unknown); Virginia Polytechnic Institute and State University (Other); William & Mary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HM20014435
Record Dates: First submitted 2019-05-09; First posted 2019-05-13 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Underage Alcohol Use; Smoking, Non-Tobacco Products
MeSH Terms: conditions — Underage Drinking; Smoking, Non-Tobacco Products

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): GMIT
  Interventions: Behavioral: GMIT
- Intervention (Experimental): Modified GMIT + Parenting support groups
  Interventions: Behavioral: GMIT+

INTERVENTIONS:
Behavioral: GMIT — Six 30-minute sessions delivered virtually in a group format. Each week a group facilitator will elicit adolescents' feedback on important topics related to substance use and provide experiential activities to help adolescents explore their beliefs and practice making healthy choices.
  Arms: Control
Behavioral: GMIT+ — Six 30-minute sessions delivered virtually in a group format. Each week a group facilitator will elicit adolescents' feedback on important topics related to substance use and provide experiential activities to help adolescents explore their beliefs and practice making healthy choices. Parents and/or guardians will virtually participate in parent-only support group sessions.
  Arms: Intervention

SUMMARY:
The purpose of this study is to compare two versions of an intervention focused on teaching 10-14-year-old Latina/o adolescent's skills that will decrease the likelihood that they will use tobacco, alcohol, and other drugs. We are also interested in determining how cultural context is related to substance use and whether additional information about other tobacco products should be added to the GMIT intervention.

DETAILED DESCRIPTION:
All adolescents will receive the Group Motivational Interviewing for Teens (GMIT) intervention. GMIT is an evidence-based group intervention that has been shown to prevent substance use among adolescents. In this project, GMIT will be delivered virtually in a group setting to multiple Latina/o adolescents. In addition, some parents will virtually participate in a parent-only support group; the other parents will not participate in any group.

In this study, participants will be randomly assigned (like flipping a coin) to receive one of two versions of an alcohol, drug, and tobacco program. As part of the program teen participants will virtually attend six 30-min intervention sessions with other teens. Parents may also participate in virtual group sessions. Participants will be asked on three separate occasions (before, immediately after, and 3 months after the sessions) to complete forms (phone/online) that ask questions about teens behavior at home, school, and in the community.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents must be between 10 and 16 years of age - parents can be any age
* Parent and adolescent must consent/assent to participate as dyad
* Self-identify as Latina/o or Hispanic

Exclusion Criteria:

* Under the age of 10 or over the age of 16
* Parent or adolescent refuses
* Identify as non-Latina/o or non-Hispanic

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 59 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2021-09-21 (Actual); Study Completion 2021-09-21 (Actual)

PRIMARY OUTCOMES:
Change in tobacco use intentions | Baseline to 3 months
  4-item self-reported tobacco use scale. Each item is scored from 1 (definitely yes) to 4 (definitely no) yielding a range between 4 and 16
Change in tobacco use attitudes | Baseline to 3 months
  7-item self-reported attitudes about tobacco scale. Each item is scored from 1 (strongly disagree) to 4 (strongly agree) yielding a range between 7 and 28
Change in smoking refusal intentions | Baseline to 3 months
  7 item self-reported smoking refusal intentions scale. Each item is scored from 1 (Definitely would say "No") to 5 (Definitely would not say "No") yielding a range from 7 to 35
Change in marijuana or other drug refusal intentions | Baseline to 3 months
  5-item self-reported marijuana or other drug refusal intentions scale. Each item is scored from 1 (Definitely would) to 5 (Definitely would not) yielding a range from 5 to 25.
Change in parent-child communication about tobacco | Baseline to 3 months
  6-item self-reported antismoking socialization scale. Item scores vary depending on response type (Yes/no or Likert scale). Total scores range from 0 to 9
Change in parental monitoring - adolescent | Baseline to 3 months
  24-item self-reported parenting practices scale completed by adolescents. Each item is scored from 1 (high monitoring) to 5 (low monitoring) yielding a range from 24 to 120
Change in parental monitoring - parent | Baseline to 3 months
  24-item self-reported parenting practices scale completed by parents. Each item is scored from 1 (high monitoring) to 5 (low monitoring) yielding a range from 24 to 120
Change in parent-child conflict - adolescent | Baseline to 3 months
  3-item conflict scale completed by adolescents. Each item is scored 1 (Never or Hardly at all) to 5 (Always or Extremely much) yielding scores ranging from 3 to 15
Change in parent-child conflict - parent | Baseline to 3 months
  20-item conflict scale completed by parents. Each item is scored 0 (False) or 1 (True) yielding scores ranging from 0 to 20
Change in family cohesiveness - adolescent | Baseline to 3 months
  10-item Family Adaptability and Cohesion Evaluation Scale completed by adolescents. Each item is scored from 1 (almost never) to 5 (almost always) yielding a range from 10 to 50.
Change in family cohesiveness - parent | Baseline to 3 months
  10-item Family Adaptability and Cohesion Evaluation Scale completed by parents. Each item is scored from 1 (almost never) to 5 (almost always) yielding a range from 10 to 50.
Change in parent-child communication - adolescent | Baseline to 3 months
  20-item Parent-Adolescent Communication Scale completed by adolescents. Each item is scored from 1 (strongly disagree) to 4 (strongly agree) yielding a range between 20 and 100.
Change in parent-child communication - parent | Baseline to 3 months
  20-item Parent-Adolescent Communication Scale completed by parents. Each item is scored from 1 (strongly disagree) to 4 (strongly agree) yielding a range between 20 and 100.

SECONDARY OUTCOMES:
Program feasibility | Baseline to 6 weeks
  Change in number of dyads enrolled in the study and number who completed the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Rosalie Corona, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No